CLINICAL TRIAL: NCT00598364
Title: Molecular Markers in the Diagnostic and Prognostic Evaluation of Thyroid Cancer
Brief Title: Molecular Markers in Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: OHSUeIRB2844
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Thyroid Cancer
Keywords: thyroid; nodule; genetic; mutation; malignancy
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thyroidectomy or neck dissection: Patients with thyroid cancer or benign thyroid disease (nodules or goiter) who underwent thyroidectomy and/or neck dissection as standard of care.

SUMMARY:
The purpose of this study is to evaluate how common gene mutations are in benign and malignant thyroid lesions.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the prevalence of molecular markers in patients with benign and malignant thyroid lesions. This study consists of:

Retrospective review of archived surgical pathology specimens at Oregon Health & Science University (OHSU) from patients with thyroid cancer or benign thyroid disease (nodules or goiter) who underwent thyroidectomy and/or neck dissection as standard of care. Molecular markers will be evaluated on archived tissue.

Molecular markers will be correlated with clinical information extracted from OHSU medical records: histologic subtype of cancer, measures of tumor aggressiveness (capsular and angiolymphatic invasion, local invasion, lymph node and distant metastases, TNM stage(TNM Classification of Malignant Tumours)) and clinical outcome (recurrence, distant metastases and death).

Patients with other malignancies presenting for standard of care services will have peripheral blood collected for DNA, RNA and buffy coat/white blood cells as a "positive" control for the DNA/RNA isolation techniques and mutation assays, as other cancers commonly express some of the same mutations. Normals will have peripheral blood collected for DNA, RNA and buffy coat/white blood cells as a "negative" control for the DNA/RNA isolation techniques and mutation assays.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 - 100
* Benign or malignant thyroid lesion, other malignancy or no thyroid abnormality
* Pathologic specimen available for analysis
* Ability to provide informed consent (for prospective study, Part Two)
* Age greater than age 18 (for normal controls)

Exclusion Criteria:

* Patients without adequate data for analysis
* Histopathologic or cytopathologic diagnosis of for medullary thyroid carcinoma (not derived from the thyroid follicular epithelium), thyroid lymphoma
* Unwilling to participate or unable to provide informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with thyroid cancer or benign thyroid disease (nodules or goiter) who underwent thyroidectomy and/or neck dissection as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 847 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is histologic lesion (benign (Graves, Hashimoto's, follicular adenoma or subtype of malignant lesion). | 7 years

SECONDARY OUTCOMES:
The main secondary outcome to be measured in malignant lesions includes measures of biologic behavior of malignant lesions including capsular and angiolymphatic invasion, local invasion and lymph node metastases at presentation | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G. Schuff, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States